CLINICAL TRIAL: NCT01693419
Title: A Phase II Study of S-1 in Combination With Gemcitabine and Erlotinib in Patients With Advanced or Metastatic Pancreatic Cancer
Brief Title: S-1, Gemcitabine and Erlotinib for Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hallym University Medical Center (Other)
Collaborators: Jeil Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMC-HO-GI-1201
Record Dates: First submitted 2012-09-20; First posted 2012-09-26 (Estimated); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Pancreas Neoplasms
Keywords: pancreas neoplasm; gemcitabine; erlotinib; S-1
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Erlotinib Hydrochloride; S 1 (combination); titanium silicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GES (Gemcitabine, Erlotinib, S-1) (Experimental): Treatment will be delivered as a 3-week cycle.
  1. Gemcitabine 1000 mg/m² IV on day 1, 8
  2. Erlotinib 100 mg/day PO on day 1
  3. S-1 60 mg/m²/day PO on day 1-14
  Interventions: Drug: GES (Gemcitabine, Erlotinib, S-1)

INTERVENTIONS:
Drug: GES (Gemcitabine, Erlotinib, S-1) — Treatment will be delivered as a 3-week cycle.
  1. Gemcitabine 1000 mg/m² IV on day 1, 8
  2. Erlotinib 100 mg/day PO on day 1
  3. S-1 60 mg/m²/day PO on day 1-14
  Other Names: Gemzar; Tarceva; TS-1

SUMMARY:
This study will conduct a phase II study of gemcitabine, erlotinib, and S-1 as first-line chemotherapy in patients with advanced pancreatic cancer and evaluate the EGFR expression, KRAS mutation, and BRAF mutation as predictive or prognostic markers

DETAILED DESCRIPTION:
Pancreatic ductal adenocarcinoma, also known as pancreatic cancer, is an eighth cause of cancer-related deaths in the world. The estimated worldwide incidence of pancreatic cancer was 277,000 cases and an estimated 266,000 patients died from the disease in 20081.

Pancreatic cancer is more common in elderly persons than in younger persons, and characterised by early locoregional spread and distant metastasis. As a result, less than 20% of patients are diagnosed with localized, potentially curable disease, and the median survival is no longer than 3-4 months without effective treatment2.

Single-agent chemotherapy with gemcitabine was considered as standard of care for patients with advanced pancreatic cancer, since Burris et al. demonstrated superiority of gemcitabine over 5-fluorouracil (5-FU) in respect of a survival benefit as well as an improvement in disease related symptoms in a randomized study3.

Nevertheless, the activity of gemcitabine monotherapy in pancreatic cancer was modest, and there was a clear need to improve its efficacy by combining it with other anticancer drugs.

Multiple agents such as 5-FU4, capecitabine5,6, cisplatin7,8, oxaliplatin9, pemetrexed10, irinotecan11, cetuximab12, and bevacizumab13, in combination with gemcitabine have been tested in clinical trials, however, they have failed to improve the outcome.

The only agent that, in combination with gemcitabine, has shown a small, but statistically significant improvement, with a hazard ratio (HR) of 0.82, the absolute improvement in median overall survival (OS) of 5.9 months with gemcitabine versus 6.2 months with the combination, is erlotinib, a small-molecule inhibitor of the epidermal growth factor receptor (EGFR)14. Considering the modest improvement in survival by adding erlotinib to gemcitabine, new combination therapy that have a great impact is urgently needed.

S-1 is an oral fluoropyrimidine derivative that combines tegafur (FT) with two modulators; 5-chloro-2, 4-dihydroxypyridine (CDHP) and oteracil potassium (Oxo) in a 1:0.4:1 molar concentration ratio. The phase II trials of a combination of gemcitabine and S-1 have demonstrated objective response rates of 32-48% and median survival of 8-12 months 15-17.

Therefore, we will conduct a phase II study of gemcitabine, erlotinib, and S-1 as first-line chemotherapy in patients with advanced pancreatic cancer and evaluate the EGFR expression, KRAS mutation, and BRAF mutation as predictive or prognostic markers.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed locally advanced unresectable, recurrent or metastatic adenocarcinoma of pancreas (Stage III-IV ; TNM staging system)
* Measurable or evaluable disease by RECIST criteria 1.1
* Minimum age of 18 years
* ECOG Performance status 0-1
* Prior adjuvant chemotherapy without gemcitabine, erlotinib or S-1 is allowed if more than 4 weeks elapsed since completion of chemotherapy.
* More than 4 weeks since completion of prior radiotherapy (measurable or evaluable lesions should be outside the radiation field)
* Adequate organ functions
* Patients must sign an informed consent indicating that they are aware of the investigational nature of the study in keeping with the policy of the hospital.

Exclusion Criteria:

* Patients treated previously with gemcitabine, erlotinib, or S-1 as adjuvant chemotherapy.
* Patients with CNS metastases
* Patients with active infection, severe heart disease, uncontrollable hypertension or diabetes mellitus, myocardial infarction during the preceding 6 months, pregnancy, or breast feeding
* Any previous or concurrent malignancy other than non-melanoma skin cancer or in situ cancer of uterine cervix
* Known history of cerebral or leptomeningeal metastases or neurologic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2011-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Objective response rate | 1.5 years
  Objective response rate will be measured from the rate of complete response (disappearance of disease) and partial response (decrease at least 30% in the sum of the longest diameters of target lesions) by RECIST (response evaluation criteria in solid tumors) guidelines.

SECONDARY OUTCOMES:
Progression free survival | 1.5 years
  Progression free survival time will be measured from the start of study treatment until documented tumor progression, or death due to any cause
Overall survival | 1.5 years
  Overall survival time will be measured from the start of study treatment until death due to any cause
Disease control rate | 1.5 years
  Disease control rate will be measured from the rate of complete response (disappearance of disease), partial response (decrease at least 30% in the sum of the longest diameters of target lesions), and stable disease (neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD) by RECIST (response evaluation criteria in solid tumors) guidelines.
Toxicity profiles | 1.5 years
  Adverse events will be descripted and graded using NCI-CTCAE version 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Dae Young Zang, DM, PhD, Principal Investigator — Hallym University Medical Center
Locations (1):
- Hallym University Medical Center, Anyang, South Korea

IPD SHARING:
Plan to Share IPD: Undecided